CLINICAL TRIAL: NCT02342587
Title: Safety and Clinical Activity of Lapatinib in Patients With HER2-positive Refractory Advanced Cancer: A Phase II Single Arm Prospective Study
Brief Title: Safety and Clinical Activity of Lapatinib in Patients With HER2-positive Refractory Advanced Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyun Lee, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-10-028
Record Dates: First submitted 2015-01-15; First posted 2015-01-21 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: HER2-positive Refractory Advanced Cancer
Keywords: Lapatinib
MeSH Terms: interventions — Lapatinib

ARMS (1):
- single arm (Experimental): Patients will be treated with oral lapatinib 1250mg once daily for 21 days.
  Interventions: Drug: Lapatinib

INTERVENTIONS:
Drug: Lapatinib — Patients will be treated with oral lapatinib 1250mg once daily for 21 days.

SUMMARY:
Although anti-HER2 (human epidermal growth factor receptor 2) therapy is currently approved for breast, gastric, and gastroesophageal cancers overexpressing the HER2 protein or amplified for the HER2 gene, HER2 aberrations (gene amplification, gene mutations, and protein overexpression) are reported in other diverse malignancies. Indeed, about 1-37% of tumors of the following types harbor HER2 aberrations: bladder, cervix, colon, endometrium, germ cell, glioblastoma, head and neck, liver, lung, ovarian, pancreas, and salivary duct.

Lapatinib is an orally active, reversible, small molecule TKI that potently inhibits both ErbB1 and ErbB2 tyrosine kinase activity. Data suggest that a dual ErbB1 and ErbB2 inhibitor may provide improved therapeutic benefit compared with inhibitors that target only one or the other receptor.

Therefore, this phase 2 study is designed to evaluated the activity of lapatinib in patients with HER2-positive refractory cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age > 19
* Written informed consent
* ECOG 0-2,
* Histologically confirmed HER2-positive Refractory solid tumor(IHC 3+ alone, or IHC 2+ with FISH amplification) and/or specific sensitivity to Lapatinib by Avatar scan that has progressed following standard therapy or that has not responded to standard therapy or for which there is no standard therapy.
* The presence of measurable disease as defined by the Response (Evaluation Criteria in Solid Tumors (RECIST) version 1.1)
* Adequate organ function

Exclusion Criteria:

* Uncontrolled symptomatic brain metastasis,Uncontrolled active infection
* Uncontrolled systemic illness (DM, CHF, unstable angina, hypertension or arrhythmia)
* Prolonged QT interval in ECG (QTc >450 msec)
* Pregnant, lactating women
* Prior treatment with lapatinib,Malabsorption syndrome, any disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, or persons unable to swallow oral medication
* Prior history of malignancy within 5 years from study entry except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer, well-treated thyroid cancer

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-12-03 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-08-21 (Actual)

PRIMARY OUTCOMES:
overall response rate | 4 weeks after treatment of lapatinib

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea